CLINICAL TRIAL: NCT03577158
Title: SAFE-AP: Automatic Control of Blood Glucose Under Announced and Unannounced Exercise
Acronym: SAFE-AP3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: Universitat Politècnica de València (Other); Universitat de Girona (Other)
Responsible Party: Principal Investigator, Ignacio Conget, Head of Endocrinology and Nutrition Department, Principal Investigator, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: SAFE-AP3
Record Dates: First submitted 2018-06-22; First posted 2018-07-05 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Diabetes Mellitus, Type 1; Insulin; Exercise; Closed-loop; Artificial Pancreas
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Insulin Resistance; Motor Activity

STUDY DESIGN:
Intervention Model Description: Longitudinal, prospective, interventional study.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Closed-loop controller with exercise mitigation module (Experimental): Sliding Mode Reference Conditioning (SMRC) Closed-loop insulin administration with mitigation module.
  Automated insulin infusion based on subcutaneous continuous glucose monitoring (CGM). Commercially available insulin infusion systems and CGM devices will be used. However, insulin infusion will be driven by the software under investigation (SAFEAP with mitigation module) based on blood glucose estimations from CGM.
  Interventions: Device: Closed-loop controller with exercise mitigation module; Device: Closed-loop controller without exercise mitigation module; Device: Open-loop insulin infusion system
- Closed-loop controller without exercise mitigation module (Experimental): Sliding Mode Reference Conditioning (SMRC) Closed-loop insulin administration. Automated insulin infusion based on subcutaneous continuous glucose monitoring (CGM). Commercially available insulin infusion systems and CGM devices will be used. However, insulin infusion will be driven by the software under investigation (SAFEAP without mitigation module) based on blood glucose estimations from CGM.
  Interventions: Device: Closed-loop controller with exercise mitigation module; Device: Closed-loop controller without exercise mitigation module; Device: Open-loop insulin infusion system
- Open-loop insulin infusion system (Active Comparator): Standard Open-loop intensive insulin treatment with continuous subcutaneous insulin infusion (CSII). Commercially available insulin infusion systems will be used.
  Interventions: Device: Closed-loop controller with exercise mitigation module; Device: Closed-loop controller without exercise mitigation module; Device: Open-loop insulin infusion system

INTERVENTIONS:
Device: Closed-loop controller with exercise mitigation module — Each subject will undergo three exercise tests, each one at 1-2 week intervals, thus completing the 3 experiments in about 6 weeks. The day of the experiment, the participant will do 3 sets of 15 minutes of cycloergometer at 70% of VO2max with 5 minutes of rest between them. On the first arm, participants will receive Sliding Mode Reference Conditioning (SMRC) Closed-loop insulin administration with a mitigation mode, based on subcutaneous continuous glucose monitoring (First arm, Closed-loop study with mitigation module).
  Commercial insulin infusion systems and continuous glucose monitoring devices will be used.
Device: Closed-loop controller without exercise mitigation module — On the second arm, participants will receive Sliding Mode Reference Conditioning (SMRC) Closed-loop insulin administration without a mitigation mode, based on subcutaneous continuous glucose monitoring (Second arm, Closed-loop study without mitigation module).
  Commercial insulin infusion systems and continuous glucose monitoring devices will be used.
Device: Open-loop insulin infusion system — Standard subcutaneous insulin infusion based on the individual insulin sensibility. Commercial insulin infusion systems and continuous subcutaneous glucose monitoring devices will be used.

SUMMARY:
Achieving near-normoglycemia has been established as the main objective for most patients with diabetes. Despite growing evidence about the health benefits of regular exercise in diabetes, exercise-associated glycemic imbalance remains a challenge in subjects with type 1 diabetes (T1D) due to a higher risk of hypoglycemia.

Automatic glucose control, the so-called artificial pancreas (AP) or closed-loop system, may represent the ideal solution for reaching the therapeutic goals in diabetic patients. Intuitively, closed-loop insulin delivery may be superior to open-loop insulin delivery due to a better compensation of the variability of subcutaneous insulin absorption and the intra-subject insulin sensitivity. However, several challenges exist to effectively realize an optimal closed-loop control of blood glucose during exercise. Indeed, the physical exercise induces one of the major glucose perturbations that need to be controlled by an artificial pancreas and is currently one of the main challenges found in clinical validations of the few existing prototypes of an artificial pancreas. In particular, experiments carried out with the currently used algorithms for glucose control (the so called PID (proportional-integrative-derivative) and MPC) showed that closed-loop insulin delivery is deteriorated by exercise, increasing the risk of hypoglycemia even with pre-exercise carbohydrate ingestion when non-announcement strategies are used.

In this project, a rigorous clinical testing of a novel closed-loop controller ('artificial pancreas') will be carried out in T1D patients treated with continuous subcutaneous insulin infusion (CSII). The innovative element of the controller is a safety auxiliary feedback based on sliding mode reference conditioning (SMRC), which has been demonstrated to limit over-insulinization and the resulting hypoglycemia, reducing glycaemic variability.

Announced and unannounced exercise will be performed in T1D subjects treated with CSII, comparing the number of hypoglycemic episodes with a controller-driven insulin delivery (closed-loop study) based on continuous subcutaneous glucose monitoring (CGM).

If any glucose value <70 mg/dL 15 gr of glucose will be provided. Moreover 15gr of glucose will be provided in AP studies when AP system recommends it.

The hypothesis is that closed loop control will provide better glycemic control, with less hypoglycemia episodes.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-65 years.
* Under CSII treatment for at least six months before visit 1.
* Body mass index between 18 and 30 kg/m2.
* HbA1c 6.0-8.5% at visit 1.
* Physical examination, laboratory data and EKG without alterations. Abnormalities considered clinically irrelevant by the investigator will not be exclusion criteria.
* Postmenopausal women or women of childbearing age using contraceptives of proven effectiveness and with negative urine pregnancy test at screening visit.

Exclusion Criteria:

* Pregnancy and breastfeeding.
* Hypoglycemia unawareness (Clarke Test >3).
* Progressive fatal disease.
* History of drug or alcohol abuse.
* History HIV positive, active hepatitis B or hepatitis C.
* Impaired liver function, as shown in, but not limited to, SGPT (serum gutamate pyruvate transaminase) or SGOT (serum glutamate oxaloacetate transaminase) more than twice the upper limit of normal at Visit 1.
* Clinically relevant microvascular complications (macroalbuminuria, pre-proliferative and proliferative retinopathy), cardiovascular, hepatic, neurological, endocrine or other systematic, apart from T1D, which may hamper the implementation of the clinical study protocol or interpretation of results study.
* Scheduled surgery during the study period.
* Mental conditions that prevent the subject to understand the nature, purpose and possible consequences of the study.
* Subjects those are unlikely to meet the clinical study protocol, eg uncooperative attitude, inability to return for follow-up visits, or poor probability of completing the study.
* Using an experimental drug or device during the past 30 days.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Number of hypoglycaemias | 180 minutes psot-exercise period
  Number of hypoglycemic episodes (defined as plasma glucose (PG) <70mg/dL) during exercise and recovery.

SECONDARY OUTCOMES:
AUC (area under curve) of PG during exercise and recovery | 180 minutes post-exercise period
  AUC0_180min, AUC0_60min and AUC60_180min of PG and time spent in different glycemic ranges (< 70; 70-180; > 180 mg/dL) during exercise and recovery.
AUC of SG during exercise and recovery | 180 minutes post-exercise period
  AUC0-180min, AUC0-60min and AUC60-180min of sensor glucose (SG) and time spent in different glycemic ranges (< 70; 70-180; > 180 mg/dL) during exercise and recovery.
Rate-of-change of glucose during exercise (ROCe) and recovery (ROCr) | 180 minutes post-exercise period

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Bondia, PhD, Study Director — Universitat Politècnica de València; Josep Vehi, PhD, Study Director — Universitat de Girona; Ignacio Conget Donlo, MD, Study Director — Hospital Clinic of Barcelona; Marga Gimenez Alvarez, MD, Study Chair — Hospital Clinic of Barcelona
Locations (1):
- Hospital Clínic de Barcelona, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Quiros C, Bertachi A, Gimenez M, Biagi L, Viaplana J, Vinals C, Vehi J, Conget I, Bondia J. Blood glucose monitoring during aerobic and anaerobic physical exercise using a new artificial pancreas system. Endocrinol Diabetes Nutr (Engl Ed). 2018 Jun-Jul;65(6):342-347. doi: 10.1016/j.endinu.2017.12.012. Epub 2018 Feb 23. English, Spanish. PMID 29483036
- [Background] Rossetti P, Quiros C, Moscardo V, Comas A, Gimenez M, Ampudia-Blasco FJ, Leon F, Montaser E, Conget I, Bondia J, Vehi J. Closed-Loop Control of Postprandial Glycemia Using an Insulin-on-Board Limitation Through Continuous Action on Glucose Target. Diabetes Technol Ther. 2017 Jun;19(6):355-362. doi: 10.1089/dia.2016.0443. Epub 2017 May 1. PMID 28459603
- [Derived] Vinals C, Beneyto A, Martin-SanJose JF, Furio-Novejarque C, Bertachi A, Bondia J, Vehi J, Conget I, Gimenez M. Artificial Pancreas With Carbohydrate Suggestion Performance for Unannounced and Announced Exercise in Type 1 Diabetes. J Clin Endocrinol Metab. 2021 Jan 1;106(1):55-63. doi: 10.1210/clinem/dgaa562. PMID 32852548